CLINICAL TRIAL: NCT03545594
Title: Traumatic Brain Injury; Needs and Treatment Options in the Chronic Phase. A Randomized Controlled Community-based Intervention
Brief Title: Traumatic Brain Injury; Needs and Treatment Options in the Chronic Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sunnaas Rehabilitation Hospital (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Cecilie Røe, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TBIcommunity
Record Dates: First submitted 2018-05-09; First posted 2018-06-04 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Traumatic Brain Injury
Keywords: Randomized trial,; Health care needs; Traumatic brain injury; Community; Goal attainment
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Independent Outcome Assessor(s) blinded to the intervention arm by masking the ID and randomization arm on the assessment and outcome forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-centered in home rehabilitation (Experimental): Eight contacts of about 2 hours duration each delivered over a 4-month period (Six in home visits and two telephone contacts before the Corona pandemic and adjusted to eight contacts and up to six of them video based when necessary during the Corona pandemic) in three phases:
  Interventions: Other: Patient-centered in home rehabilitation
- Control (Active Comparator): Usual follow-up assessment and health care and rehabilitation services provided in the municipality
  Interventions: Other: Control

INTERVENTIONS:
Other: Patient-centered in home rehabilitation — Eight contacts (six in-home visits of 1-2 hours duration each and two telephone contacts before the Corona pandemic and eight sessions with up to six of them video delivered if necessary during the Corona pandemic ) delivered over a 4-month period in three phases
  Arms: Patient-centered in home rehabilitation
Other: Control — Usual follow-up in the municipality
  Arms: Control

SUMMARY:
Traumatic brain injury (TBI) is a condition affecting the persons' central nervous system with a need for extensive and highly specialized initial health care provision followed by comprehensive rehabilitation efforts. Frequent and life-long medical, cognitive, emotional and behavioral changes are expected. The community-based services are largely responsible for dealing with the chronic challenges affecting people with TBI.

120 patients >16 years at the time of injury and between 18 and 72 years at inclusion, with clinical TBI diagnosis on acute admission and verified injury-related intracranial abnormalities reporting cognitive, emotional and physical problems more than 2 years after the injury will be included and randomized to a patient-centered in-home program intervention and treatment as usual. The intervention consists of an individualized and goal-oriented intervention will be provided in the persons' home environment, in close collaboration with family members and local health care providers when available. Assessments will be conducted at baseline, at the end of the intervention 4 months after inclusion and one year after inclusion. Primary outcome is participation (Part-O) and TBI specific health related quality of life (Qolibri). Secondary outcomes include goal attainment within individualized targeted outcome areas, depression and anxiety, symptom burden, unmet health care needs and acceptability of intervention as assessed by patient, family member and health professional. The project will contribute to increased understanding of knowledge transfer processes, and dissemination of evidence based practice for TBI. Thus, the project has the potential to improve the current health care for patients with TBI and its delivery.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a condition affecting the persons' central nervous system with a need for extensive and highly specialized initial health care provision followed by comprehensive rehabilitation efforts. Frequent and life-long medical, cognitive, emotional and behavioral changes are expected. The community-based services are largely responsible for dealing with the chronic challenges affecting people with TBI.

120 patients >16 years at the time of injury and between 18 and 72 years at inclusion, with clinical TBI diagnosis on acute admission and verified injury-related intracranial abnormalities reporting cognitive, emotional and physical problems more than 2 years after the injury will be included and randomized to a patient-centered in-home program intervention and treatment as usual. The intervention consists of individualized and goal-oriented strategies provided in the persons' home environment in close collaboration with family members and local health care providers. The original protocol describes a total of 8 sessions of which 2 will be telephone based. Due to the Corona pandemic hittting Norway in March 2020 the home visits had to be reduced and adapted to the individual situation of the participants. The protocol now includes 8 sessions with up to 6 of them being delivered by video. The intervention will be provided in addition to the usual treatment the participants receive in the municipality. The control group will receive the usual treatment provided in the municipality. Assessments will be conducted at baseline, at the end of the intervention 4-5 months after inclusion and one year after inclusion. Primary outcome is participation (Part-O) and TBI specific health related quality of life (Qolibri). Secondary outcomes include goal attainment within individualized targeted outcome areas, depression and anxiety, symptom burden, unmet health care needs and acceptability of intervention as assessed by patient, family member and health professional. In March 2020 a few additional questions regarding the impact of the Corona pandemic on health and participation has been included. The closedown periods of the Norwegian Society during Covid-19 will be used as covariate and/or predictors in the analysis. The project will contribute to increased understanding of knowledge transfer processes, and dissemination of evidence based practice for TBI. Thus, the project has the potential to improve the current health care for patients with TBI and its delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients >16 years at injury and 18-72 years at inclusion, with clinical TBI diagnosis on acute admission and CT/MRI verified injury-related intracranial abnormalities.
* Patients reporting TBI-related cognitive, emotional and physical problems and/or reduced physical and mental health and/or difficulties with participation in activities with family, friends and in the community at least 2 years after the injury,
* Able to provide informed consent and collaborate in the goal setting processing.
* Living at home at study inclusion.

Exclusion Criteria:

* Patients are excluded if they have severe preexisting neurological disorder that would confound outcome assessments and severe psychiatric diseases
* Patients unable to provide informed consent or participate in a goal-setting process.
* Participants with insufficient fluency in Norwegian to allow for communication with therapists and outcome assessors will also be excluded.
* Substance abuce or history of violence that could represent a security risk for the professionals delivering the intervention

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Participation | 12 months
  Participation assessment and Recombined Tools- Objective (PART-O) (Social domain)
General Health | 12 months
  Quality of Life after Brain Injury (Qolibri overall scale, sum score of 6 items )

SECONDARY OUTCOMES:
Global functioning | 4 and 12 months
  Glasgow outcome scale extended (GOSE) (score 0-8)
Depression | 4 months (patients and family) and 12 months intervention (patients)
  Patients Health Questionnaire (PHQ-9) (patients and family members)
Physical and mental health (EQ-5D) and quality-adjusted life years, (QALYs) | 4 and 12 months
  Physical and mental health (scored according to the EQ-5D algoritm )and QALYs (patients) and overall health (on a scale 0-100,family members)
Acceptability and satisfaction with the intervention | 4 and 12 months
  Acceptability Scale assessed by patients, care providers and family members (sum score)
Target outcome areas | 4 and 12 months
  The patient nominate their three most important problems and the difficulties they have with them on a scale from 0 to 4. Changes in the difficulty score is evaluated.
Symptom burden | 4 and 12 months
  Rivermead post-concussion questionnaire (RPQ)(patients) (scoring algoritm)
Patient and family members, evaluating self-awareness and functioning. Patient and family members, evaluating self-awareness and functioning | 4 and 12 months
  Patient Competency Rating Scale (PCRS) (sum score) rated by patient and family member
Caregiver burden (Caregiver burden scale) | 4 and 12 months
  Caregiver burden-family member
Anxiety Disorder Measurement (GAD-7) | 4 and 12 months
  Generalised Anxiety Disorder Measurement (GAD-7) (sumscore 7 items, 0-21)
Participation | 4 months
  Participation assessment and Recombined Tools- Objective (PART-O) (3 domains and total score
General Health | 4 months
  Quality of Life after Brain Injury (Qolibri overall scale, sum score of 6 items )
Participation | 12 months
  Participation assessment and Recombined Tools- Objective (PART-O) (domain Round and about and Productivity, Total score

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Røe, Study Chair — OUH
Locations (1):
- OUH, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Only aggregated data will be shared according to the Norwegian legislation

REFERENCES:
- [Derived] Lovstad M, Borgen IMH, Hauger SL, Kleffelgard I, Brunborg C, Roe C, Soberg HL, Forslund MV. Family member reported symptom burden, predictors of caregiver burden and treatment effects in a goal-oriented community-based randomized controlled trial in the chronic phase of traumatic brain injury. BMC Neurol. 2024 Sep 10;24(1):333. doi: 10.1186/s12883-024-03841-7. PMID 39256658
- [Derived] Kleffelgard I, Forslund M, Hauger S, Roe C, Bragstad LK, Soberg HL, Lovstad M, Borgen IMH. Process evaluation of a complex intervention evaluating the effectiveness of home-based rehabilitation in the chronic phase of traumatic brain injury. Disabil Rehabil. 2024 Dec;46(25):6134-6142. doi: 10.1080/09638288.2024.2324119. Epub 2024 Mar 6. PMID 38445314
- [Derived] Borgen IMH, Lovstad M, Hauger SL, Forslund MV, Kleffelgard I, Andelic N, Sveen U, Soberg HL, Sigurdardottir S, Winter L, Lindstad MO, Brunborg C, Roe C. Effect of an Individually Tailored and Home-Based Intervention in the Chronic Phase of Traumatic Brain Injury: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2310821. doi: 10.1001/jamanetworkopen.2023.10821. PMID 37145600
- [Derived] Borgen IMH, Lovstad M, Andelic N, Hauger S, Sigurdardottir S, Soberg HL, Sveen U, Forslund MV, Kleffelgard I, Lindstad MO, Winter L, Roe C. Traumatic brain injury-needs and treatment options in the chronic phase: Study protocol for a randomized controlled community-based intervention. Trials. 2020 Mar 27;21(1):294. doi: 10.1186/s13063-020-4195-5. PMID 32216840